# 知情同意书

#### 研究背景介绍:

您将被邀请参加一项,由<u>南方医科大学药学院和东莞市人民医院</u>共同主持的研究。本研究是<u>观察丹参酮胶囊治疗新型冠状病毒感染的有效性</u>,它将历时 <u>14-60 天</u>。此研究由<u>广东省防治</u>新型冠状病毒科技攻关项目资助进行。由于您是新型冠状病毒感染者而被邀请加入此项研究。

本知情同意书提供给您一些信息以帮助您决定是否参加此项研究。您参加本项研究完全是自愿的。本次研究已通过东莞市人民医院生物医学伦理审查委员会审查。

请您仔细阅读该知情同意书,有任何疑问请随时向负责该项研究的研究者提出。

# 研究目的:

新冠病毒的变异导致多国面临疫情多次暴发难题,基因突变可改变病毒的传播力、致病性、免疫原性等,如目前全世界流行的 Omicron 变异毒株传播速度更快、传染性增强、感染群体年轻化,继而影响抗病毒药物的疗效或减弱疫苗的保护效率! 因此,为充分应对新冠病毒的变异以及未来可能的新发冠状病毒,研发广谱抗冠状病毒药物是当前迫切的临床需求。丹参酮胶囊系已上市药物,采用传统中药丹参根部脂溶性成分入药,功能主治抗菌消炎,用于痤疮、扁桃腺炎、疖,其在临床上的使用缓解了抗生素耐药性和毒性大的局面。研究团队前期基础研究证明丹参酮胶囊在体外与人源化 ACE2 转基因小鼠中具有抗新冠病毒活性,使用丹参酮胶囊治疗新冠病毒感染,可进一步拓宽丹参酮胶囊抗病毒的药理活性,可能增加其作为抗病毒感染药物的临床功能主治。一方面,丹参酮胶囊为中药口服胶囊,具有生产/运输成本低、安全性高、患者依从性高等优势,另一方面,丹参酮胶囊有望在防治新冠病毒感染的同时,降低患者机体炎症水平,改善新冠病毒所致肺炎(COVID-19)症状,可较高程度满足新冠肺炎药物研发的重大需求。

本研究为扩大丹参酮胶囊临床功能主治的研究者发起的临床试验,基于新型冠状病毒肺炎抗病毒新药研究临床试验技术指导原则,拟通过纳排标准纳入新冠感染者(轻型和/或中型)160例,开展安慰剂平行对照试验,设置丹参酮胶囊干预组与丹参酮胶囊安慰剂对照组。通过测定患者核酸转阴时间/率、新冠长期后遗症发生率、血清生化等指标评价丹参酮胶囊(国药准字Z13020110)治疗新冠病毒感染的安全性与有效性。

#### 纳入标准:

- 1. 符合国家卫生健康委员会发布的《新型冠状病毒感染诊疗方案 (试行第十版)》关于新冠病毒感染的诊断,根据病原学或血清学检测,确诊 2 天内,且同时满足以下条件:
- 1) 新型冠状病毒感染核酸检测 N 基因和 ORF 基因 Ct 值均<30(荧光定量 PCR 方法,界限值为 40):
- 2) 临床分型属于轻型和/或中型:受试者在筛选时至少具有以下一个或多个症状评分≥1分的COVID-19临床症状,包括但不限于:发热,咳嗽,咽喉痛,鼻塞或者流鼻涕,头痛,肌肉痛,恶心,呕吐,腹泻,气促或者呼吸困难,畏寒或者寒战。
- 2. 年龄 18-65 岁, 性别不限;

- 3. 受试者需满足以下一项或多项: 1) 筛选期阳性 SARS-CoV-2 病毒感染测定的样本距首次给予试验用药品≤3 天, 2) 首次出现 COVID-19 症状距首次给予试验用药品≤3 天:
- 4. 患者自愿参与本研究,本人或其法定代表人签署书面知情同意书,愿意配合随访。

#### 排除标准:

- 1. 根据《新型冠状病毒感染诊疗方案(试行第十版)》,重症/危重症高危人群、进入研究前确诊 为重型、危重型的患者;
- 2. 在进入研究前已接受抗病毒治疗,例如接受中成药或中药方剂治疗、Paxlovid、利托那韦片、SARS-CoV-2 单克隆抗体治疗、康复者恢复期血浆、其他以新型冠状感染为适应症的临床试验药物等治疗(既往新冠感染治疗除外);
- 3. 已知对治疗药物丹参酮胶囊过敏及过敏体质(包括对其他药物易产生过敏反应)受试者;
- 4. 现患有严重影响免疫系统的疾病,如:人类免疫缺陷病毒(HIV)感染,或血液系统,或脾切除、器官移植术等;
- 5. 妊娠期、哺乳期女性;
- 6. 筛选期疑似有除了新冠病毒之外的细菌、真菌、病毒或其他感染;
- 7. 进入研究前患有支气管肺炎、慢性肺脓肿、慢性咳嗽 8 周以上、慢性咽喉炎伴咳嗽等疾病;
- 8. 在筛选期有下列情况之一: 1) ALT 或 AST>1.5 倍 ULN; 2) eGFR<60mL/min; 3) 血红蛋白<8.0g/L, 血小板<5000/μL;
- 9. 近3个月内参与过其他临床试验的患者;
- 10. 根据研究者的判断,不官入组者。

# 研究过程和方法:

本研究将选取共 160 例新冠肺炎患者,证明丹参酮胶囊治疗新型冠状病毒肺炎的有效性。如果您同意参与这项研究,我们将对您进行编号,建立病历档案并随机分配至干预组或安慰剂对照组。所有受试者根据《新型冠状病毒感染诊疗方案 (试行第十版)》,均接受常规的对症治疗,包括维持水/电解质平衡、高热者进行物理降温或给予解热药物、咳嗽咳痰严重者给予止咳祛痰药物。期间干预组给予丹参酮胶囊,一次 4 粒,一日 3 次,对照组给予丹参酮胶囊安慰剂,一次 4 粒,一日 3 次,随餐口服,治疗期为 5 天,停药时间取决于您临床症状消失的时间与核酸转阴的时间。研究期间您需每日定点来院,由医护人员对您进行每日一次的鼻/咽拭子采集,检测新冠病毒核酸水平;每日由医护人员指导填写一份临床症状评分表;分别于给药当天与停药当天采集您的外周血 10 毫升,监测血常规与血清炎症因子。您的样本仅用于本次研究,研究结束后将按照医学常规进行销毁,样本如涉及外送检测,我们将提前告知您并取得您的同意。停药后第 14±2 天、第 30±2 天、第 60±2 各随访一次,将收集您的鼻/口咽部样本复查核酸(根据受试者回访时的实际情况由临床医生决定是否进行)、并对您进行"新冠后遗症"症状评分与心脑血管系统检查(包括血压、心率、心肌酶、D-2 聚体、同型半胱氨酸、心电图、动态心电图、心脏彩超、脑 CT等)。

# 研究可能的获益:

本研究将为您提供免费的治疗与相关检测,通过对您的标本进行检测将有助于对疾病作出 诊断,为您的治疗提供必要的建议,您将直接获益。您的样本也为疾病的研究提供有益的信息, 有利于该疾病的防控和治疗。

治疗期间,本研究将为您提供 500 元/人/天\*(用药天数)的补贴,按照实际用药天数给予补贴(停药时间取决于您临床症状消失的时间与核酸转阴的时间),中途退出的按实际情况给予补贴,补贴将以现金的形式发放给您。

# 研究风险与不适:

研究干预措施可能产生的风险: 丹参酮胶囊不良反应包括轻度肠胃道不适包括恶心、肠胃胀气、腹部不适和腹泻, 个别人可能有过敏反应; 根据国家药品不良反应监测系统数据显示, 丹参酮胶囊累计不良反应报告率为十万分之一, 不良反应发生属于非常罕见级别的比例, 患者可耐受或停药后自行恢复。此外安慰剂胶囊可能引起轻微不适包括头痛、恶心或乏力。

您的样本采集将严格按照要求操作,标本的采集可能会有一些非常小的风险,包括在研究 进行过程中需要采集血样进行血常规、血生化等检查。血样采集可能引起短暂的疼痛、局部青 紫,针刺部位瘀斑或出血,少数人会有轻度头晕,或极为罕见的针头感染。

# 其他治疗干预方式:

除研究用药外,受试者可以合并常规对症治疗使用的药物,不允许合并使用其他中成药/中药。根据病情进展,对于发病 5 天以内的中型成年患者,我们将参照《新型冠状病毒感染诊疗方案(试行第十版)》,给予抗病毒治疗(阿兹夫定片:空腹整片吞服,每次 5mg,每日 1 次)。

# 隐私问题:

如果您决定参加本项研究,您参加试验及在试验中的个人资料均属保密。对于您来说,所有的信息将是保密的。例如:您的血标本将以研究编号数字而非您的姓名加以标识。可以识别您身份的信息将不会透露给研究小组以外的成员,除非获得您的许可。如果标识符必须保留,说明为什么。说明何时销毁(书写的或用其他方式记录的)研究资料。如果研究结束时,资料没有销毁,介绍资料保存在何处和保存多久。说明在未来将如何使用保存的资料,以及如何获得受试者允许在未来使用他们的资料。所有的研究成员和研究申办方都被要求对您的身份保密。您的档案将保存在研究机构档案柜中,仅供研究人员查阅。为确保研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅您的个人资料。

在您和其他受试者的理解和协助下,通过本项目研究的结果可能会在医学杂志上发表,但 是我们会按照法律的要求为您的研究记录保密。

# 参加研究可能涉及的花费

(说明受试者参加该研究可能涉及的花费,明确研究将支付的具体费用等。) 参与本研究将不会给您带来额外的花费。

# 研究相关损害的赔偿

如果您因参与这项研究而受到伤害:如发生与该项临床研究相关的损害时,南方医科大学将根据我国相关法律提供相应的赔偿。

#### 自由退出:

作为受试者,您可随时了解与本研究有关的信息资料和研究进展,自愿决定(继续)参加还是不(继续)参加。参加后,无论是否发生伤害,或是否严重,您可以选择在任何时候通知研究者要求退出研究,您的数据将不纳入研究结果,您的任何医疗待遇与权益不会因此而受到影响。如果继续参加研究,会对您造成严重的伤害,研究者也将会中止研究的进行。

但在参加研究期间,请您提供有关自身病史和当前身体状况的真实情况;告诉研究医生自己在本次研究期间所出现的任何不适;不得服用受限制的药物、食物等;告诉研究医生自己在最近是否曾参与其他研究,或目前正参与其他研究。如果因为您没有遵守研究计划,或者发生了与研究相关的损伤或者有任何其它原因,研究医师可以终止您继续参与本项研究。

# 联系方式:

如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本项研究相关的问题,您可以与<u>胡国栋</u>(研究者姓名)联系咨询,电话 <u>18819326682</u>。

如果您在参加研究过程中,有任何关于受试者权益相关的问题,您可以联系<u>东莞市人民医</u>院医学伦理委员会,电话:\_\_\_\_\_\_电子邮件:\_\_\_\_\_。

# 知情同意签字:

| 我已经阅读了 | 本知情同意 | 书,并且我 | 的研究人员 | l | (签字)已经 | 2.将此次研究的 |
|---|---|---|---|---|---|---|
| 目的、内容、风险 | 和受益情况 | 1向我作了详 | 羊细的解释说 | 说明,对我询 | 同的所有问题せ | 2给予了解答, |
| 我对此项研究已经 | 了解,我自 | 愿参加本项 | ī研究。我签 | 署了两份知情 | <b>青同意书,并保</b> | 存了其中一份。 |
| 受试者签名: | | | | | | |
| 日期: | | | | | | |
| (注,加里受运 | 学者不识字时 | ·冶季贝证人 | <i>数夕 加里码</i> | 过考无行为能 | 力时则需代理人 | <i>同音</i> ) |
| (江: 知本文山 | V4-1, PV 1_h1 | 4 m 兆 | <i>亚石,州木又</i> | W(11 /L1) /YHE, | / 【 4 1 火 1 冊 1 【 4 注 / 【 1 | |
| 我已经告知了 | 受试者本知 | 1情同意书的 | 的相关内容, | 并将此次研究 | 究的目的、内容<br>2000年 | 孚、风险和受益 |
| 情况向受试者作了 | 详细的解释 | 经说明,对受 | ·<br>运者询问的 | 的所有问题也给 | <b>给予了解答。</b> 受 | を试者签署了两 |
| 份知情同意书,并 | 留存了其中 | 一份。 | | | | |
| 研究者签名: | | | | | | |
| 日期: | | ——<br>Н | | | | |
| | <del>_</del> | / ] | $\vdash$ | | | |